CLINICAL TRIAL: NCT02535156
Title: Schizotypal Personality Disorder Risperidone
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: CIM/02/112/01
Record Dates: First submitted 2015-08-22; First posted 2015-08-28 (Estimated); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Schizotypal Personality Disorder
MeSH Terms: conditions — Schizotypal Personality Disorder | interventions — Risperidone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Schizotypal Personality Disorder (Experimental): Schizotypal Personality Disorder (SPD) patients. They received two interventions: risperidone 1 mg and placebo (lactose).
  Interventions: Drug: Risperidone; Drug: Placebo
- Healthy controls (Experimental): Control group consisting of healthy volunteers.They received two interventions: risperidone 1 mg and placebo (lactose).
  Interventions: Drug: Risperidone; Drug: Placebo

INTERVENTIONS:
Drug: Risperidone — 1 mg Risperidone
Drug: Placebo — Lactose Placebo

SUMMARY:
Neurophysiological indices of self-monitoring were assessed in a group of patients with Schizotypal Personality Disorder (SPD) and a control group. Both groups were assessed after the administration of risperidone and placebo.

DETAILED DESCRIPTION:
The electroencephalogram (EEG) was recorder while participants (SPD participants and controls) performed a behavioral task: the Eriksen Flanker Task. The continuous EEG was segmented, corrected for artifacts and averaged. A component of the event-related brain potential known as the error-related negativity (ERN) was identified and its amplitude quantified in microvolts.

This procedure was conducted two hours after the administration of risperidone 1 mg and placebo (lactose) on two different experimental days and for each participant group (SPD patients and controls).

The amplitude of the ERN after placebo was compared between groups to test for baseline (non-drug-induced) differences between patients and controls.

The impact of risperidone on the amplitude of the ERN was compared between the two participant groups.

ELIGIBILITY:
Inclusion Criteria:

* Schizotypal Personality Disorder

Exclusion Criteria:

* Major Psychiatric Disorder
* Medical condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2003-01; Primary Completion 2014-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Neurophysiological indices of self-monitoring (Error Related Negativity) | During acute effects of pharmacological treatment (up to 2 hours)
  Amplitude of the Error Related Negativity was assessed prior to and 2 hours after treatment administration